CLINICAL TRIAL: NCT04994574
Title: Effects of Tiotropium/Olodaterol on Cardio-pulmonary Exercise Capacity in Patients With Hyperinflated Chronic Obstructive Pulmonary Disease [ACHIEVE]
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-0635
Record Dates: First submitted 2021-07-12; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tiotropium/olodaterol (Experimental)
  Interventions: Drug: tiotropium/olodaterol

INTERVENTIONS:
Drug: tiotropium/olodaterol — From Visit 2(Baseline), test subjects will be use tiotropium/olodaterol inhaler once a day for 4 weeks. After that, visit the hospital at 4 weeks to receive examination and terminate participation.

SUMMARY:
[Background] Hyperinflation caused by increased airflow limitation and emphysema change commonly accompanies dyspnea, which leads to inactivity, reducing exercise capacity, and deconditioning. Hyperinflation in COPD is also associated with decreased left and right end-diastolic volume and stroke volume, and cardiac output.

Previous studies investigated effects of ICS/LABA or LABA/LAMA versus placebo on cardiac function in patients with COPD and lung hyperinflation. However, there are not evidences for effects of LABA/LAMA on cardio-pulmonary exercise capacity.

Cardiopulmonary exercise testing (CPET) is an exercise stress test with concomitant expired gas analysis, which provides objective parameters of functional capacity. Since CPET can assess integrated exercise responses of cardiopulmonary, vascular, and skeletomuscular systems, it can reveal abnormalities that are not apparent in a resting state. Moreover, change in oxygen consumption during exercise and anaerobic threshold can be evaluated.

The investigators would like to investigate change in cardio-pulmonary exercise capacity via CPET before and after tiotropium/olodaterol inhalation in COPD patients with hyperinflation, which is the first clinical study. Association between change in cardio-pulmonary exercise capacity with function of heart and lung would be further evaluated with cardiac magnetic resonance (CMR) and lung function.

The in investigators expect to enhance cardio-pulmonary exercise capacity though the improvement in cardiac and pulmonary function with tiotropium/olodaterol inhalation. This result would provide evidence to encourage to treat with dual bronchodilators in COPD patients with hyperinflation.

[Study objectives] To investigate and compare the bronchodilator effect of tiotropium/olodaterol on cardio-pulmonary exercise capacity in hyperinflated COPD patients

[Study design] Prospective, single-center, one-arm clinical study After using the tiotropium/olodaterol inhaler for 4weeks, the investigators will compare pre- and post- cardio-pulmonary exercise capacity, cardiac function, lung function, symptoms and quality of life

[Statistic methods] For continuous variables, data will be presented as median, minimum, maximum with standard deviation (95% confidence intervals). For categorical variables, data will be presented as percentage (95% confidence intervals). Paired t-test for continuous variables and chi-squared test for categorical variables will be performed to compare the difference in results before and after inhalation of the tiotropium/olodaterol inhaler.

This is a pilot study; therefore, sample size cannot be calculated by power analysis, because of the absence of any data in the literature that could be reviewed. A sample size is expected to be 40 patients. When the drop-out rate 10% is considered, final sample size is expected to be 44.

ELIGIBILITY:
Inclusion Criteria:

1. The person who voluntarily signed the consent form
2. Adults over 40 years of age
3. Patients who diagnosed with COPD
4. Patients with smoking history of 10 packs or more
5. Patients who are taking or in need of tiotropium/olodaterol inhaler for the treatment of COPD
6. Patients in a clinically stable state within 3 months of screening
7. Patients who confirmed FEV1/FVC < 0.7 and FEV1 <80% after using bronchodilator
8. Patients who confirmed FRC > 125%
9. Patients who confirmed mMRC > 2

Exclusion Criteria:

1. Patients with a history of asthma
2. Patients with asthma- COPD overlap
3. Patients with serious disease other than COPD
4. Patients with unstable or life-threatening cardiac arrhythmias
5. Patients hospitalized for heart failure or myocardial infarction within 1 year of screening
6. Patients with systolic ejection fraction less than 40%
7. Patients with unstable ischemic heart disease
8. Patients receiving regular oxygen therapy for 1hour or more per day
9. Others who are difficult to participate in the research under judgment of the investigation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Change of maximum oxygen consumption | At 4 weeks
  After 4 weeks of tiotropium/olodaterol inhaler use, measure the change in the maximum oxygen consumption (VO2, ml/kg/min) during the cardio-pulmonary exercise test compared to the baseline

SECONDARY OUTCOMES:
Change in cardiopulmonary exercise test results after 4 weeks compared to baseline | At 4 weeks
  After 4 weeks of tiotropium/olodaterol inhaler use, measure the secondary outcomes during the cardio-pulmonary exercise test compared to the baseline
Change in cardiac MRI results after 4 weeks compared to baseline | At 4 weeks
  After 4 weeks of tiotropium/olodaterol inhaler use, measure the secondary outcomes during the cardiac MR compared to the baseline
Change in echocardiography results after 4 weeks compared to baseline | At 4 weeks
  After 4 weeks of tiotropium/olodaterol inhaler use, measure the secondary outcomes during the echocardiography compared to the baseline
Change in spirometry results after 4 weeks compared to baseline | At 4 weeks
  After 4 weeks of tiotropium/olodaterol inhaler use, measure the secondary outcomes during pulmonary function test compared to the baseline
Change in questionnaire evaluation and quality of life (CAT score) after 4 weeks compared to baseline | At 4 weeks
  < Questionnaire >
  COPD Assessment Test(CAT) score : from 0 to 40, the higher scores denote a more severe impact of COPD on patient's life
Change in questionnaire evaluation and quality of life (mMRC score) after 4 weeks compared to baseline | At 4 weeks
  < Questionnaire >
  Modified Medical Research Council(mMRC) scale : from 0 to 4, the higher scale, the more deterioration in severity of dyspnea
Change in questionnaire evaluation and quality of life (BDI score) after 4 weeks compared to baseline | At 4 weeks
  < Questionnaire >
  Baseline Dyspnea Index(BDI score : from 0 to 12, the lower the score, the more deterioration in severity of dyspnea
Change in questionnaire evaluation and quality of life (TDI score) after 4 weeks compared to baseline | At 4 weeks
  < Questionnaire >
  Transitional Dyspnea Index(TDI) score : from -9 to +9, the lower the score, the more deterioration in severity of dyspnea
Change in serologic cardiac biomarkers after 4 weeks compared to baseline | At 4 weeks
  < Serologic cardiac biomarker>
  NTproBNP, high sensitive troponin, soluble ST2

CONTACTS AND LOCATIONS:
Overall Officials: Ji Ye Jung, Principal Investigator — Severance Hospital, Yonsei University Health System
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cazzola M, Rogliani P, Matera MG. Cardiovascular disease in patients with COPD. Lancet Respir Med. 2015 Aug;3(8):593-5. doi: 10.1016/S2213-2600(15)00279-9. Epub 2015 Jul 22. No abstract available. PMID 26208993
- [Background] de Miguel Diez J, Chancafe Morgan J, Jimenez Garcia R. The association between COPD and heart failure risk: a review. Int J Chron Obstruct Pulmon Dis. 2013;8:305-12. doi: 10.2147/COPD.S31236. Epub 2013 Jun 28. PMID 23847414
- [Background] Kessler R, Partridge MR, Miravitlles M, Cazzola M, Vogelmeier C, Leynaud D, Ostinelli J. Symptom variability in patients with severe COPD: a pan-European cross-sectional study. Eur Respir J. 2011 Feb;37(2):264-72. doi: 10.1183/09031936.00051110. Epub 2010 Nov 29. PMID 21115606
- [Background] Labaki WW, Xia M, Murray S, Curtis JL, Barr RG, Bhatt SP, Bleecker ER, Hansel NN, Cooper CB, Dransfield MT, Wells JM, Hoffman EA, Kanner RE, Paine R 3rd, Ortega VE, Peters SP, Krishnan JA, Bowler RP, Couper DJ, Woodruff PG, Martinez FJ, Martinez CH, Han MK. NT-proBNP in stable COPD and future exacerbation risk: Analysis of the SPIROMICS cohort. Respir Med. 2018 Jul;140:87-93. doi: 10.1016/j.rmed.2018.06.005. Epub 2018 Jun 5. PMID 29957287
- [Background] Ledwidge M, Gallagher J, Conlon C, Tallon E, O'Connell E, Dawkins I, Watson C, O'Hanlon R, Bermingham M, Patle A, Badabhagni MR, Murtagh G, Voon V, Tilson L, Barry M, McDonald L, Maurer B, McDonald K. Natriuretic peptide-based screening and collaborative care for heart failure: the STOP-HF randomized trial. JAMA. 2013 Jul 3;310(1):66-74. doi: 10.1001/jama.2013.7588. PMID 23821090
- [Background] Ledwidge MT, O'Connell E, Gallagher J, Tilson L, James S, Voon V, Bermingham M, Tallon E, Watson C, O'Hanlon R, Barry M, McDonald K. Cost-effectiveness of natriuretic peptide-based screening and collaborative care: a report from the STOP-HF (St Vincent's Screening TO Prevent Heart Failure) study. Eur J Heart Fail. 2015 Jul;17(7):672-9. doi: 10.1002/ejhf.286. PMID 26139583